CLINICAL TRIAL: NCT03185091
Title: Safety of Rapid Ventricular Pacing During Cerebral Aneurysm Surgery by Multimodal Neuromonitoring
Brief Title: Neuromonitoring During Rapid Ventricular Pacing in Patients Undergoing Cerebral Aneurysm Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, ethisch.comite@uza.be, Principal Investigator, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 12/50/410
Record Dates: First submitted 2015-06-24; First posted 2017-06-14 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Arterial Aneurysm; Ventricular Rate Response Pacing
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rapid ventricular pacing (Other): Safety of rapid ventricular pacing during neurosurgical procedures
  Interventions: Other: rapid ventricular pacing; Procedure: Surgery

INTERVENTIONS:
Other: rapid ventricular pacing
Procedure: Surgery

SUMMARY:
To evaluate the effect of rapid ventricular pacing on the oxygenation of the brain in patients scheduled for cerebral aneurysm clipping surgery or arteriovenous malformation surgery.

DETAILED DESCRIPTION:
Patients scheduled for cerebral aneurysm clipping surgery or arteriovenous malformation surgery(ASA 1to 3 over 18years) receive standard care general anesthesia including central venous line for rapid ventricular pacing technique. A contralateral Foresight sensor is placed on the forehead of the patient at induction. After the craniotomy two micro electrodes(PBtO2 and cerebral blood flow) are placed in the brain and fixated. A subdural strip electrode is placed on the surface of the brain to record the electrical activity. Effect of mild hyperventilation and oxygenation with 100% O2 is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for cerebral aneurysm surgery or arterial venous malformation
* American Society of Anesthesiologists classification 1, 2, or 3

Exclusion Criteria:

* non

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-01-14 (Actual); Primary Completion 2016-04-11 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Cerebral oxygenation during surgery | During surgery
  Oxygenation of the brain is measured by near-infrared spectroscopy and by evaluation of the brain tissue oxygen pressure by two microelectrodes placed in the brain.
Cerebral blood flow during surgery | During surgery
  Thermal diffusion flowmetry measures the local absolute cerebral blood flow

SECONDARY OUTCOMES:
Electrophysiological changes in the brain during surgery | During surgery
  Electro-corticography measures electrophysiological changes in the brain.
Effect of ventilation with 100 % oxygen on cerebral parameters after rapid ventricular pacing | Intraoperative ( Start of ventilation at 100% oxygen until bloodgas analyses shows an increase in arterial oxygen pressure.)
  Effect of ventilation with 100% oxygen on cerebral blood flow and cerebral tissue oxygenation measured by thermal diffusion flowmetry and brain tissue oxygen pressure measured by microelectrodes placed in the brain in combination with near-infrared spectroscopy, respectively.
Effect of hyperventilation on cerebral parameters after rapid ventricular pacing | Intraoperative (Start of hyperventilation until bloodgas analyses shows an arterial carbon dioxide pressure between 24 and 32 millimetre of mercury.)
  Effect of hyperventilation (defined as arterial carbon dioxide pressure between 24 and 32 millimeter mercury) on cerebral blood flow and cerebral tissue oxygenation measured by thermal diffusion flowmetry and brain tissue oxygen pressure measured by microelectrodes placed in the brain in combination with near-infrared spectroscopy, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Vera Saldien, MD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Saldien V, Menovsky T, Rommens M, Van der Steen G, Van Loock K, Vermeersch G, Mott C, Bosmans J, De Ridder D, Maas AI. Rapid ventricular pacing for flow arrest during cerebrovascular surgery: revival of an old concept. Neurosurgery. 2012 Jun;70(2 Suppl Operative):270-5. doi: 10.1227/NEU.0b013e318236d84a. PMID 21937926